CLINICAL TRIAL: NCT02790151
Title: Memory Rehabilitation by Means of Working Memory Training in Combination
Brief Title: Memory Rehabilitation by Means of Working Memory Training in Combination With a Recollection Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oldenburg (Other)
Responsible Party: Principal Investigator, Kim Merle Richter, MSc Psychologie, University of Oldenburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UOLDENBURG
Record Dates: First submitted 2015-03-02; First posted 2016-06-03 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Memory Deficits
Keywords: working memory, recollection training, transfer
MeSH Terms: conditions — Memory Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy (Active Comparator): Learning and practicing memory strategies
  Interventions: Behavioral: Standard Therapy
- Experimental Intervention (Experimental): Computerbased working memory training and Recollection training
  Interventions: Behavioral: Experimental Intervention

INTERVENTIONS:
Behavioral: Standard Therapy — Learning and practicing Memory strategies
  Arms: Standard Therapy
Behavioral: Experimental Intervention — Computerbased Working Memory Training in Combination with a Recollection Training
  Arms: Experimental Intervention

SUMMARY:
Memory deficits after brain damage are common and there is still a need for evaluated therapy methods. In this study we compare two therapeutic interventions and investigate whether therapy effects can be found on neuropsychological tests and on a test measuring memory in everyday life.

DETAILED DESCRIPTION:
In the interventiongroup a computerbased working memory training is combined with a recollection training (repitition-lag procedure). The patients in the active control group undergo the standard memory therapy that is normally provided in the rehabilitation centre (with a focus on the acquisition and execution of different memory strategies, e.g. the spaced retrieval method). The patients in both groups are tested on different neuropsychological tests before and after nine hours of therapy. Additionally, a test is conducted that assesses memory in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* brain injury
* memory deficits (performance below average in the California Verbal Learning Test in learning trial 1 or 5, sfr or lfr)

Exclusion Criteria:

* severe amnesia (less than 2 words in sfr of the CVLT), dementia, sensory or motor aphasia, impaired vision, insufficient German language skills, lack of patient's consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Test to assess change in memory performance in everyday life | baseline and 9 hours
  The test includes different single tasks that measure memory in everyday life e.g. Story recall (Subtest 6 from the Rivermead Behavioral Memory Test) Outcome measure: Total number of points

SECONDARY OUTCOMES:
Outcome change in different neuropsychological tests | baseline and 9 hours
  Tests for verbal memory, working memory, prospective memory, attention and word fluency (Composite scores built from raw scores)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Hildebrandt, Prof. Dr., Study Director — Universität Oldenburg
Locations (1):
- Rehabilitationszentrum GmbH, Oldenburg, Deutschland, Germany

REFERENCES:
- [Derived] Richter KM, Modden C, Eling P, Hildebrandt H. Improving everyday memory performance after acquired brain injury: An RCT on recollection and working memory training. Neuropsychology. 2018 Jul;32(5):586-596. doi: 10.1037/neu0000445. Epub 2018 Apr 26. PMID 29697993